CLINICAL TRIAL: NCT02522923
Title: Comparison of Two Different Initial Entry Portals of Care for Patients Seeking Care for Musculoskeletal Pain: A Multisite Randomized Controlled Trial
Brief Title: Back-on-Track Studying Early Quality Care
Acronym: on-Track
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Temple University (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23131
Record Dates: First submitted 2015-07-29; First posted 2015-08-13 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Musculoskeletal Diseases
Keywords: Physical Therapy Modalities; Primary Care; Health Services Research
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Physical Therapists; Physicians, Primary Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapist (Experimental): Participants randomized to this arm will receive care from a physical therapist first.
  Interventions: Other: Physical Therapist
- Primary Care Provider (Active Comparator): Participants randomized to this arm will receive care from a primary care provider first.
  Interventions: Other: Primary Care Provider

INTERVENTIONS:
Other: Physical Therapist — The participant will receive an evaluation and intervention from a physical therapist. The patient will be referred onward to other providers as needed.
  Arms: Physical Therapist
Other: Primary Care Provider — The participant will receive an evaluation and intervention from a primary care provider. The patient will be referred onward to other providers as needed.
  Arms: Primary Care Provider

SUMMARY:
This study is a randomized controlled trial conducted at two clinical sites. The purpose of this study is to determine whether patients with musculoskeletal injuries do better by seeing a primary care provider first versus seeing a physical therapist first. Target enrollment is 150 subjects.

DETAILED DESCRIPTION:
Physical therapists have an important role as initial contact providers for individuals with musculoskeletal disorders. Health care expenditures are on the rise each year in the U.S. and a large proportion is due to musculoskeletal disorders. Despite the rise in spending, there has not been an improvement in outcomes for individuals with musculoskeletal disorders. Furthermore, increased medical spending and utilization could expose patients to iatrogenic harm. Comparative effectiveness studies of different portals of entry would help to determine the most effective pathways for individuals with musculoskeletal disorders to seek care. The purpose of this study is to determine whether patients with musculoskeletal injuries do better by seeing a primary care provider first versus seeing a physical therapist first. Subjects will be enrolled from two sites (Temple University, Philadelphia, PA and Brooke Army Medical Center, San Antonio, TX). Patient self-reported outcomes measures will be collected at baseline and 6 weeks. At 6 months, healthcare utilization will be assessed. The investigators plan to enroll a target sample size of 75 subjects per site (150 total). Descriptive statistics will be computed to characterize the 2 treatment groups with ANCOVA being used to assess differences between treatment groups at 6 weeks, adjusting for baseline values, evaluating the assumption of parallel slopes. The investigators will further investigate sources of systematic differences in response to treatment using methods such as generalized estimating equations and linear mixed effects models. This research will be the first multi-site study to compare effectiveness of these two pathways for individuals with musculoskeletal pain in the U.S. With a growing older adult population, the percentage of individuals who have musculoskeletal pain in the U.S. will only increase over time. This research study is timely and could meet the need for identifying the most effective pathway for individuals with musculoskeletal pain to seek care.

ELIGIBILITY:
Inclusion Criteria:

1. A patient at Temple University Employee Health, OR, Brooke Army Medical Center.
2. Able to speak English sufficiently to understand informed consent
3. A patient with a musculoskeletal condition as their primary complaint
4. Greater than 18 years old
5. Within 90 days (3 months) of either initial musculoskeletal onset or repeat acute recurrence of a previous episode

Exclusion Criteria:

1. Patients have already sought care from provider for their presenting condition for this current episode
2. Patients have an insurance plan that requires them to see an outside provider prior to seeing the study providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Physical function on the 10-item short form PROMIS global health measure | 6 weeks

SECONDARY OUTCOMES:
Physical function on the Patient Specific Functional Scale | 6 weeks
Overall Improvement on the Global Rating of Change | 6 weeks
Patient Satisfaction on a Likert scale | 6 weeks
Acceptability of Symptom State on the PASS | 6 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 weeks
Percentage of Subjects using Over-the-counter or Prescription Medication to Assess Medication Usage | 6 weeks
Number of Limited or Light Duty Days to Measure Work Status | 6 weeks
Number of Physical Therapy or Medical Appointments or Tests orders as a Measure of Health care utilization | 6 months
Presenteeism as Measured by Participation at Work on Likert Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heidi A Ojha, D.P.T., Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Temple University Employee Health, Philadelphia, Pennsylvania
  - Brooke Army Medical Center, Fort Sam Houston, Texas

REFERENCES:
- [Result] Moore JH, McMillian DJ, Rosenthal MD, Weishaar MD. Risk determination for patients with direct access to physical therapy in military health care facilities. J Orthop Sports Phys Ther. 2005 Oct;35(10):674-8. doi: 10.2519/jospt.2005.35.10.674. PMID 16294989